CLINICAL TRIAL: NCT03645005
Title: An e-Health Intervention to Improve Symptom Burden and Health-Related Quality of Life Among Hispanic Women Completing Active Treatment for Breast Cancer
Brief Title: A Research Study for Latina Women After Breast Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Betina Yanez, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00201961
Record Dates: First submitted 2018-04-24; First posted 2018-08-24 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Cancer-related Problem/Condition; Quality of Life; Stress, Emotional
Keywords: eHealth; Health Related Quality of Life; Symptom Burden; Breast Cancer; Hispanic
MeSH Terms: conditions — Stress, Psychological; Breast Neoplasms | interventions — Self-Management

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- My Guide (psychoeducation & self-management program) (Experimental)
  Interventions: Behavioral: "My Guide" (psychoeducation & self-management program)
- My Health (health education program) (Active Comparator)
  Interventions: Behavioral: "My Health" (health education program)

INTERVENTIONS:
Behavioral: "My Guide" (psychoeducation & self-management program) — "My Guide" is a Smartphone application incorporating elements informed by the extant literature, designed to improve quality of life and symptom burden among Hispanic breast cancer survivors. "My Guide" components are designed to improve breast cancer knowledge, cancer-relevant self-efficacy, stress and symptom management skills, Both intervention and active comparator conditions are administered to participants for 8 weeks.
  Arms: My Guide (psychoeducation & self-management program)
Behavioral: "My Health" (health education program) — "My Health" is a health promotion Smartphone application with health education content on nutrition, and general advice on lifestyle choices and prevention. The "My Health" control content was based on similar content tested in other psychosocial interventions with cancer survivors. Both intervention and active comparator conditions are administered to participants for 8 weeks.
  Arms: My Health (health education program)

SUMMARY:
The purpose of this study is to examine the effects of a developed psychosocial eHealth intervention on the proposed primary outcomes, health-related quality of life and symptom burden, among Hispanic breast cancer survivors.

The intervention components include breast cancer knowledge, stress awareness and management, social support, and enhanced communication and intimacy skills. The intervention will be delivered via a Smartphone application over an 8-week period.

Participants are randomized into either an intervention application (described above) or a control application (health information and health promotion strategies). Aside from using the Smartphone application for the recommended 8 weeks, participation in this study includes three assessments: baseline (at the beginning of the research study), 6-week follow-up, and 8-week follow-up.

DETAILED DESCRIPTION:
Among Hispanics, the largest and fastest growing ethnic minority group in the U.S., cancer is the leading cause of death whereas cardiovascular disease is the leading cause of death for African Americans and non-Hispanic Whites (NHWs). Hispanics also experience substantially lower rates of 5-year cancer-specific survival relative to non-Hispanic Whites (NHWs). Hispanic cancer patients in the U.S. also report significantly worse cancer-related symptom burden and health-related quality of life (HRQOL) than NHWs, even after adjusting for socioeconomic factors. Despite this, very few randomized, intervention studies have specifically targeted cancer-related symptom burden and HRQOL outcomes among Hispanic women, especially during the period at the end of active treatment which is a critical period to intervene to provide skills and tools to assist with this transition. Innovative approaches to providing interventions such as Smartphone technology are especially important for this patient population. Ubiquitous Smartphone use among ethnic minorities in the US provide a unique opportunity to implement a pragmatic technology- and evidence-based psychosocial intervention that overcomes some access to care barriers as well as time and logistical constraints. Furthermore, given that Hispanics own Smartphones and seek health information online from a mobile device at similar or higher rates than other groups in the U.S., Smartphone interventions offer an opportunity to overcome obstacles to accessing resources and services that can be culturally informed and provide skills to improve symptom burden and HRQOL. This study aims to create and evaluate a culturally informed eHealth psychoeducational and psychosocial intervention for English or Spanish-speaking Hispanic women completing treatment for breast cancer. This intervention is grounded in evidence-based paradigms to improve the proposed Primary Outcomes: Cancer-Related Symptom Burden and HRQOL and the proposed Secondary Outcomes: usability and markers the intervention use. This study is designed in two-phases to develop and test a Smartphone-based intervention that can be disseminated to cancer survivors at a relatively low cost. The first phase is intended to create an eHealth intervention designed to improve cancer-related symptom burden and HRQOL. The second phase is designed as an 8-week randomized trial intended to evaluate the eHealth intervention when compared to a control condition. It is hypothesized that the eHealth intervention will significantly improve cancer-related symptom burden and HRQOL compared to the control condition.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Diagnosis of breast cancer, non-metastatic, stage 0-IIIA; for women diagnosed with stage 0, either radiation or chemotherapy is required as an additional treatment to surgery
3. Completed active treatment for breast cancer (surgery, chemotherapy and/or radiation therapy, current hormonal treatment allowed)
4. No current evidence of disease
5. Within 3 to 24 months post-active treatment [e.g., surgery, chemotherapy, radiation, or combination of the two or three]
6. at least 21 years of age
7. Able to speak and read English or Spanish
8. Able to provide informed consent
9. Elevated score on breast cancer symptom burden and HRQoL, measured by the Functional Assessment of Cancer Therapy-Breast using an established cut-off score for clinically meaningful, compromised HRQoL
10. Self-identified Hispanic/Latina ethnicity.

Exclusion Criteria:

1. Visual, hearing, voice, or motor impairment that would prevent completion of study procedures
2. diagnosis of an unmanaged psychotic disorder, bipolar disorder, dissociative disorder, or other diagnosis for which participation in this trial is either inappropriate or dangerous - this includes patients who have life-threatening illness (e.g., end-stage kidney disease) or diagnosis of a chronic disease that is associated with a major functional impairment (e.g., fibromyalgia)
3. Illicit substance or alcohol dependence
4. Suicidal ideation, plan, intent
5. Alzheimer's, dementia or history of stroke
6. Scheduled reconstruction surgery within 1 month of any study procedures or involvement.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life will be evaluated with The Functional Assessment of Cancer Therapy-Breast (FACT-B) | HRQoL will be first assessed at baseline (T1), initial HRQoL changes will be assessed at 6 weeks post-baseline (T2), and finally any additional HRQoL changes will be captured 8 weeks post-baseline (T3)
  The FACT-B has been used extensively to measure HRQoL, and has been translated to and validated in Spanish. The FACT-B assesses participant's wellbeing in physical, emotional, social, functional, and breast cancer related concerns in the last seven days using a five-point response scale.
Symptom Burden will be evaluated with The Breast Cancer Prevention Trial symptom questionnaire (BCPT) | Symptom Burden will be first assessed at baseline (T1), initial changes will be assessed at 6 weeks post-baseline (T2), and finally any additional changes will be captured 8 weeks post-baseline (T3)
  The BCPT measures participants' symptom burden. The BCPT asks participants to report their level of discomfort with 25 breast cancer related symptoms during the past four weeks using a five-point response scale.

SECONDARY OUTCOMES:
Cancer-Specific Distress will be evaluated using The Impact of Event Scale (IES) | Cancer-Specific Distress will be first assessed at baseline (T1), initial changes will be assessed at 6 weeks post-baseline (T2), and finally any additional changes will be captured 8 weeks post-baseline (T3)
  The IES is made up of two subscales measuring the frequency of intrusion and avoidance experiences after a stressful event. The IES has been widely used among patients diagnosed with cancer and has been translated and validated with Spanish-speaking participants.
Breast Cancer Related Knowledge will be evaluated with the Knowledge about Breast Cancer Questionnaire | Breast Cancer Knowledge will be first assessed at baseline (T1), initial changes will be assessed at 6 weeks post-baseline (T2), and finally any additional changes will be captured 8 weeks post-baseline (T3)
  This questionnaire has been tested with Spanish-speaking Hispanic breast cancer survivors, it is made up of 16 true and false questions regarding general breast cancer knowledge.
Breast Cancer Related Communication and Attitudinal Self-Efficacy will be evaluated using the Communication and Attitudinal Self-Efficacy scale for cancer (CASE-cancer) | Breast Cancer Related Communication and Attitudinal Self-Efficacy will be first assessed at baseline (T1), initial changes will be assessed at 6 weeks post-baseline (T2), and finally any additional changes will be captured 8 weeks post-baseline (T3)
  The CASE-cancer questionnaire is made up various subscales measuring breast cancer related communication and attitudinal self-efficacy. Each question asks participants to use a four-point response scale to agree or disagree with statements regarding their level of confidence with different skills.
Stress Management Skills will be evaluated with the Brief COPE Inventory | Stress Management Skills will be first assessed at baseline (T1), initial changes will be assessed at 6 weeks post-baseline (T2), and finally any additional changes will be captured 8 weeks post-baseline (T3)
  The Brief COPE is made up of various subscales measuring different ways of coping. Each question as participants to rate how often they have used each coping mechanism in response to their breast cancer experience.

CONTACTS AND LOCATIONS:
Overall Officials: Betina Yanez, Ph.D., Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - University of Illinois Cancer Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baik SH, Oswald LB, Buscemi J, Buitrago D, Iacobelli F, Perez-Tamayo A, Guitelman J, Penedo FJ, Yanez B. Patterns of Use of Smartphone-Based Interventions Among Latina Breast Cancer Survivors: Secondary Analysis of a Pilot Randomized Controlled Trial. JMIR Cancer. 2020 Dec 8;6(2):e17538. doi: 10.2196/17538. PMID 33289669

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT03645005/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT03645005/ICF_001.pdf